CLINICAL TRIAL: NCT01851083
Title: A Phase 2 Multicenter Trial of Pediatric Autologous Bone Marrow Mononuclear Cells (BMMNCs) for Severe Traumatic Brain Injury (TBI)
Brief Title: Pediatric Autologous Bone Marrow Mononuclear Cells for Severe Traumatic Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Charles Cox, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-13-0038; R01NS077963 (NIH)
Record Dates: First submitted 2013-05-05; First posted 2013-05-10 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; TBI; pediatric; acute; stem cells
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- autologous bone marrow mononuclear cells (Experimental): a bone marrow harvest will be performed, followed by a single intravenous infusion of autologous bone marrow mononuclear cells within 48 hours of injury.
  Interventions: Biological: autologous bone marrow mononuclear cells
- placebo infusion (Placebo Comparator): a sham harvest will be performed, followed by a single intravenous placebo infusion within 48 hours of injury.
  Interventions: Other: Placebo Infusion

INTERVENTIONS:
Biological: autologous bone marrow mononuclear cells — BMMNC infusion of either 6x10^6 cells/kg or 10x10^6 cells/kg weight.
  Other Names: BMMNCs
  Arms: autologous bone marrow mononuclear cells
Other: Placebo Infusion — Placebo infusion of 0.9% Sodium Chloride
  Other Names: Saline Infusion
  Arms: placebo infusion

SUMMARY:
Pediatric severe traumatic brain injury (TBI) is the leading cause of death and disability in children ages 1-14 years old. There are no effective therapies to treat secondary brain injury and the post-injury response of CNS apoptosis and neuroinflammation. This study is a follow-up trial from a previously performed Phase I trial that demonstrated the safety and potential CNS structural preservation effect of intravenous autologous bone marrow mononuclear cells (BMMNC) after severe TBI in children. (Cox, 2011) The study is designed as a prospective, randomized, placebo controlled, blinded Phase 2 safety/biological activity study. The investigators hope to determine the effect of intravenous infusion of autologous BMMNCs on brain structure and neurocognitive/functional outcomes after severe TBI in children.

DETAILED DESCRIPTION:
Study Design: Multicenter, randomized, blinded, placebo controlled, Bayesian adaptive dose escalation design.

Study Intervention: Single dose administered within 48 hours from time of injury. Controls will undergo a sham harvest and receive similarly labeled/external appearance and volume of 0.9% NaCl. BMMNC's will be harvested and undergo processing under cGMP conditions to obtain 6x10^6 cells/kg or 10x10^6 cells/kg weight. The cellular product/placebo will be infused within 48 hours of injury.

Safety Monitoring & Follow-Up: Subjects will be monitored for infusion related toxicity post-infusion through hospital discharge and follow-up return study visits. Laboratory and imaging studies will be repeated at the 1, 6, and 12-month follow-up visits. A medical safety monitor (MSM) will review blinded SAE reports following post-infusion Day 14 for each subject in real time to ensure good clinical practice and to quickly identify safety concerns. The MSM will remain blinded to the treatment assignment, unless the NINDS appointed DSMB approves unblinding.

ELIGIBILITY:
Inclusion Criteria:

1. Between 5 and 17 years of age on the day of injury,
2. Glasgow Coma Score (GCS) between 3 and 8, (best un-medicated post-resuscitation score during screening),
3. Ability to obtain legally authorized representative (LAR) consent, and complete the BMMNC/Sham harvest and cell/placebo infusion within 48 hours of the initial injury,
4. Ability to speak English or Spanish.

Exclusion Criteria:

1. Known history of: a. previous brain injury, b. intellectual deficiency or psychiatric condition, defined as inability to independently function in a regular classroom that may invalidate our ability to assess post-injury changes in cognition or behavior (ADHD and/or other learning disabilities are NOT an exclusion), c. neurologic impairment and/or deficit, d. seizure disorder requiring anti-convulsant therapy, e. recently treated infection, f. renal disease or altered renal function (post-resuscitation serum creatinine > 1.5 mg/dL), g. hepatic disease or altered liver function (post-resuscitation, non-contusion related SGPT > 150 μ/L and/or T. Bilirubin >1.3 mg/dL), h. cancer, i. immunosuppression as defined by WBC < 3, 000 cells/ml at admission, j. HIV+, k. chemical or ETOH dependency, l. history of child abuse, m. premature birth (<37 weeks GA/2500 grams) resulting in cognitive/physical disabilities and/or developmental delay.
2. Obliteration of perimesencephalic cistern on initial head CT/MRI suggesting prolonged hypoxic ischemic insult/herniation syndrome.
3. Initial hospital ICP > 40 mm Hg.
4. Hemodynamic instability at the time of screening defined as SBP <90 mmHg, ongoing fluid resuscitation and/or requirement for inotropic support to maintain MAP at or above normal for age - does not include CPP based inotropic support. IVF alone does not exclude from enrollment.
5. Uncorrected coagulopathy at the time of bone marrow harvest defined as INR > 1.6, PTT > 38 sec; PLT< 100,000; Fibrinogen < 100 g/dL.
6. Unstable pelvic fractures defined as requiring early operative fixation.
7. Pulmonary contusions defined as a chest x-ray with non-anatomic opacification and/or PaO2:FiO2 ratio < 250 associated with the mechanism of injury.
8. Greater than AAST Grade 3 solid or hollow visceral injury of the abdomen and/or pelvis as diagnosed by CT or other imaging.
9. Spinal cord injury diagnosed by CT/MR imaging or clinical findings.
10. Persistent hypoxia defined as SaO2 < 94% for > 30 minutes occurring at any time from hospital admission to time of consent.
11. Positive pregnancy test, if applicable.
12. Concurrent participation in an interventional drug/device research study.
13. Unwillingness to return for follow-up visits.
14. Contraindications to MRI.
15. Penetrating brain injury.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2013-08; Primary Completion 2020-09-16 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
brain white matter and gray matter structural preservation on diffusion tensor magnetic resonance imaging (DTMRI) | one year post infusion
  DTMRI quantitative indices of both macro and microscopic integrity will be evaluated and compared to DTMRI of immediate post-injury treated and non-treated controls.

SECONDARY OUTCOMES:
CNS white matter and gray matter preservation in regions of interest and improves functional and neurocognitive deficits in children after TBI | one year post infusion

OTHER OUTCOMES:
Infusional toxicity safety evaluations | 7 days post-infusion
  Murray Score and liver function tests

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Cox, Jr., M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Phoenix Children's Hospital I University of Arizona, Phoenix, Arizona
  - The University of Texas Health Science Center at Houston, Houston, Texas